CLINICAL TRIAL: NCT02992275
Title: Neuromuscular Electrical Stimulation as an Adjunct to Improve Hip Abductor Muscle Quality and Reduce Fall Risk
Brief Title: NMES to Improve Hip Abductor Strength and Balance
Acronym: IMAGINE+NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Odessa Addison, Research Scientist, Baltimore VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00072630
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postural Balance
Keywords: Hip; Muscle; Skeletal/physiopathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMES + MMBI (Experimental): Neuromuscular electrical stimulation applied to hip abductors along with participation in a multi-modality balance intervention
  Interventions: Other: Neuromuscular electrical stimulation (NMES); Other: Multi-Modality Balance Intervention (MMBI)

INTERVENTIONS:
Other: Neuromuscular electrical stimulation (NMES) — Participants will receive NMES to the hip abductors while performing strength training 3 times per week for 24 weeks
Other: Multi-Modality Balance Intervention (MMBI) — Participants will attend a group balance class that focuses on movement and obstacle negotiation 3 times per week for 24 weeks

SUMMARY:
This study will examine the addition of neuromuscular electrical stimulation (NMES) on the hip abductors during strength training and a fall prevention program for improving muscle strength and improving balance. All individuals in this study will receive NMES to their hip abductors and will participate in a fall reduction program.

DETAILED DESCRIPTION:
Falls are a leading cause of disability in older adults. Decreased lower extremity muscle mass and strength contribute to balance and mobility limitations. Our more recent work also suggests that in addition to the traditional targets of muscle mass of the thigh and leg muscles, dysfunction of the hip abductors may contribute to balance and mobility limitations resulting in increased fall risk. Older adults with impaired hip abductor muscles demonstrate increased amounts of intramuscular fat (IMAT) in and around the muscles, decreased hip abductor strength, lower balance scores, increased gait variability (a predictor of future falls), and poor stepping mechanics when recovering from a balance perturbation. Increased IMAT and muscle dysfunction of the hip abductors may contribute to poor hip abductor muscle recruitment and make changing these muscle during a traditional intervention difficult. Neuromuscular electrical stimulation (NMES) is one method to improve muscle mass, strength and quality in older adults, but has not traditionally been used on the hip abductors. We propose that a targeted multimodality balance intervention (MMBI) focused on the lateral and diagonal stepping and hip abductor strengthening when combined with NMES will result in improvements in mobility and balance.

ELIGIBILITY:
Inclusion Criteria:

Mobility and balance limitations as demonstrated by a self-reported fall within the past year or requiring greater than 8 seconds to complete the 4-square step test

-

Exclusion Criteria:

1. Cardiovascular Risks: Poorly controlled hypertension (>160/100); or patient report of: symptomatic angina at rest or during exercise, syncope without known resolution of cause, or a significant coronary event (such as a MI) in the past six months
2. COPD requiring home oxygen
3. Contraindications to resistance training, including a self-reported history of intracranial or retinal bleeding in the last year or Diabetes with active proliferative retinopathy
4. Patient report of significant spinal stenosis that would limit participation in the exercise intervention
5. Non-ambulatory mobility status or a transtibial or transfemoral amputation
6. Dementia (on medical record review or mini-mental status exam score <24).
7. Other severe medical illness or condition that would preclude safe participation in the study as determined by the study team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mobility | 6 months
  Mobility will be measured with the use of the mini-BesTest

SECONDARY OUTCOMES:
Balance | 6-months
  Balance will be measured with the four-square step test
Muscle Strength | 6-months
  Muscle strength will be measured as hip abductor strength quantified by use of a biodex

CONTACTS AND LOCATIONS:
Overall Officials: Les Katzel, MD, PhD, Study Director — Director Baltmore GRECC; Odessa Addison, DPT, PhD, Principal Investigator — Research Scientist
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No